CLINICAL TRIAL: NCT03281538
Title: An Open-Label, Multicenter, Extension Study to Evaluate the Long Term Safety of Intravenous CR845 in Hemodialysis Patients With Chronic Kidney Disease-Associated Pruritus
Brief Title: Extension Study to Evaluate IV CR845 in Hemodialysis Patients With Moderate-to-Severe Pruritus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR845-CLIN3101
Record Dates: First submitted 2017-06-20; First posted 2017-09-13 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Uremic Pruritus
Keywords: CR845; difelikefalin; Pruritus; Chronic Itch; Itch; Itching; hemodialysis; Uremic Pruritus; Dialysis; CKD; CKD-associated pruritus; CKD-aP; ESRD (end stage renal disease); Chronic Kidney Disease; Kidney failure, chronic; Kidney dysfunction; Generalized pruritus
MeSH Terms: conditions — Pruritus; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CR845 0.5mcg/kg (Experimental): CR845 0.5mcg/kg IV medication administered three times/week after dialysis
  Interventions: Drug: CR845

INTERVENTIONS:
Drug: CR845 — IV CR845 0.5 mcg/kg administered after each dialysis session (3 times/week)

SUMMARY:
This is an open-label multicenter, long-term extension safety study to evaluate the safety of IV CR845 administered after each dialysis session over a Treatment Period of up to 52 weeks.

DETAILED DESCRIPTION:
This is an open-label multicenter, long-term extension safety study to evaluate the safety of IV CR845 administered after each dialysis session over a Treatment Period of up to 52 weeks. This study will consist of a Screening Visit, a 52 week Treatment Period, and a Follow-up Visit. Informed consent will be obtained prior to performing any study-specific procedures. All patients will have a Screening Visit, which can be performed anytime within 14 days prior to the first dose of study drug, to confirm eligibility.

Clinical laboratory tests, electrocardiograms (ECGs), vital signs, adverse events, and concomitant medications will be monitored throughout the study. Blood samples for inflammatory biomarkers will be collected from all patients prior to dialysis on Day 1 and periodically until the End of Treatment or Early Termination Visit. Blood samples will also be collected periodically for clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

1. Willing and able to provide written informed consent prior to participating in this study;
2. Able to communicate clearly with the Investigator and staff, able to understand the study procedures, and able and willing to comply with the study schedules and all study requirements;
3. Males or females 18 years of age or older;
4. Currently on hemodialysis for end-stage renal disease and has been categorized as experiencing moderate to severe uremic pruritus;
5. If female:

   1. Is not of childbearing potential (surgically sterile or postmenopausal, as defined in Section 6.5.1.6); or
   2. Has a negative serum pregnancy test at screening and agrees to use acceptable contraceptive measures (as defined in Section 6.5.1.6) from the time of informed consent until the safety Follow-up Visit or 7 days after the last dose of study drug, whichever is later.
6. If male, agrees not to donate sperm after the first dose of study drug until 7 days after the last dose, and agrees to use a condom with spermicide or abstain from heterosexual intercourse during the study until 7 days after study drug administration. (Note: No restrictions are required for a vasectomized male provided his vasectomy was performed ≥4 months prior to dosing);
7. Has a dry body weight of ≥40.0 kg at screening (prescription target dry body weight);
8. Has adequacy of dialysis, defined as meeting 1 of the following criteria during the 3 months prior to screening:

   1. ≥2 single pool Kt/V measurements ≥1.2; or
   2. ≥2 urea reduction ratio measurements ≥65%; or
   3. 1 single pool Kt/V measurement ≥1.2 and 1 urea reduction ratio measurement ≥65%

Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

1. Received an investigational drugwithin 30 days prior to the first dose of study drug, or is planning to participate in another interventional clinical study while enrolled in this study.
2. Has a concomitant disease or any medical condition that, in the opinion of the Investigator, could pose undue risk to the patient, impede completion of the study procedures, or would compromise the validity of the study measurements, including, but not limited to:

   1. Known or suspected history of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, -diagnosed alcohol, narcotic or other drug abuse, or substance dependence within 12 months prior to screening;
   2. New York Heart Association Class IV congestive heart failure (Appendix 1, Section 14.0);
   3. Severe mental illness or cognitive impairment (eg, dementia);
   4. Any other relevant acute or chronic medical or neuropsychiatric condition;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederique Menzaghi, Study Director — Cara Therapeutics
Locations (25):
- United States (24):
  - Cara Therapeutics Study Site, Chula Vista, California
  - Cara Therapeutics Study Site, El Centro, California
  - Cara Therapeutics Study Site, Long Beach, California
  - Cara Therapeutics Study Site, Northridge, California
  - Cara Therapeutics Study Site, Denver, Colorado
  - Cara Therapeutics Study Site, Hollywood, Florida
  - Cara Therapeutics Study Site, Tampa, Florida
  - Cara Therapeutics Study Site, Winter Park, Florida
  - Cara Therapeutics Study Site, Albany, Georgia
  - Cara Therapeutics Study Site, Augusta, Georgia
  - Cara Therapeutics Study Site, Meridian, Idaho
  - Cara Therapeutics Study Site, Springfield, Massachusetts
  - Cara Therapeutics Study Site, Roseville, Michigan
  - Cara Therapeutics Study Site, Kansas City, Missouri
  - Cara Therapeutics Study Site, Albuquerque, New Mexico
  - Cara Therapeutics Study Site, Gallup, New Mexico
  - Cara Therapeutics Study Site, Mineola, New York
  - Cara Therapeutics Study Site, Ridgewood, New York
  - Cara Therapeutics Study Site, Bethlehem, Pennsylvania
  - Cara Therapeutics Study Site, Knoxville, Tennessee
  - Cara Therapeutics Study Site, El Paso, Texas
  - Cara Therapeutics Study Site, San Antonio, Texas
  - Cara Therapeutics Study Site, St. George, Utah
  - Cara Therapeutics Study Site, Wauwatosa, Wisconsin
- Cara Therapeutics Study Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fishbane S, Wen W, Munera C, Lin R, Bagal S, McCafferty K, Menzaghi F, Goncalves J. Safety and Tolerability of Difelikefalin for the Treatment of Moderate to Severe Pruritus in Hemodialysis Patients: Pooled Analysis From the Phase 3 Clinical Trial Program. Kidney Med. 2022 Jun 28;4(8):100513. doi: 10.1016/j.xkme.2022.100513. eCollection 2022 Aug. PMID 36039153

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CR845 0.5mcg/kg
Started | 288
Completed | 133
Not Completed | 155

BASELINE CHARACTERISTICS:
Arm/Group | CR845 0.5mcg/kg
Number analyzed (Participants) | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 173
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 148
  White | 114
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With AEs
Description: Assessed by physical examination, monitoring of adverse events, vital signs and laboratory assessments
Time Frame: Up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CR845 0.5mcg/kg
Number analyzed (Participants) | 288
Participants | 240

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Arm/Group | CR845 0.5mcg/kg
All-Cause Mortality (participants affected / at risk) | 17/288
Serious Adverse Events (participants affected / at risk) | 148/288
Other Adverse Events (participants affected / at risk) | 139/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 0.5mcg/kg (N=288)
Anaemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 14
Angina pectoris (Cardiac disorders) | 8
Cardiac arrest (Cardiac disorders) | 8
Cardiac failure congestive (Cardiac disorders) | 8
Atrial fibrillation (Cardiac disorders) | 4
Coronary artery disease (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 3
Mitral valve incompetence (Cardiac disorders) | 2
Acute left ventricular failure (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Chronic left ventricular failure (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardia ischaemia (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Diplopia (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Discoloured vomit (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 8
Asthenia (General disorders) | 4
Death (General disorders) | 2
Impaired healing (General disorders) | 2
Catheter site thrombosis (General disorders) | 1
Chest pain (General disorders) | 1
Complication associated with device (General disorders) | 1
Drug interaction (General disorders) | 1
Sudden death (General disorders) | 1
Vascular stent restenosis (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 12
Sepsis (Infections and infestations) | 9
Bacteraemia (Infections and infestations) | 6
Cellulitis (Infections and infestations) | 6
Osteomyelitis (Infections and infestations) | 5
Clostridium difficile colitis (Infections and infestations) | 3
Gangrene (Infections and infestations) | 3
Septic shock (Infections and infestations) | 3
Infected skin ulcer (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Ateriovenous fistula site infection (Infections and infestations) | 1
Ateriovenous graft site abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Cardiac valve vegetation (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Latent tuberculosis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1
Serratia sepsis (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Subacute endocarditis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Vascular access site infection (Infections and infestations) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 3
Vascular access malfunction (Injury, poisoning and procedural complications) | 3
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 2
Abdominal injury (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1
Chemical burn of respiratory tract (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Skin wound (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1
Blood pressure increased (Investigations) | 1
Cardiac stress test abnormal (Investigations) | 1
Electrocardiogram T wave inversion (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2
Calciphylaxis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Bening lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 3
Brain stem infarction (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 2
Brain injury (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Hypertensive encephalopathy (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Unresponsive to stimuli (Nervous system disorders) | 1
Device expulsion (Product Issues) | 1
Mental status changes (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Genital lesion (Reproductive system and breast disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia apsiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 9
Hypertensive emergency (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 2
Shock haemorrhagic (Vascular disorders) | 2
Steal syndrome (Vascular disorders) | 2
Accelerated hypertension (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Arterial stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Peripheral venous disease (Vascular disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Shunt thrombosis (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CR845 0.5mcg/kg (N=288)
Nausea (Gastrointestinal disorders) | 48
Diarrhoea (Gastrointestinal disorders) | 44
Fall (Injury, poisoning and procedural complications) | 42
Vomiting (Gastrointestinal disorders) | 38
Hypotension (Vascular disorders) | 30
Non-cardiac chest pain (General disorders) | 22
Dizziness (Nervous system disorders) | 21
Abdominal pain (Gastrointestinal disorders) | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT03281538/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT03281538/SAP_001.pdf